CLINICAL TRIAL: NCT01039649
Title: Quantifying Radiation Induced Changes in Pulmonary Function in Irradiated and Non-irradiated Lung Tissue
Brief Title: A Study to Test Lung Function After Radiation Therapy
Acronym: PFS
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, John M. Buatti, Professor and Chair, Radiation Oncology, University of Iowa
Other Study IDs: 200905703
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Lung Neoplasms; Neoplasm Metastasis
Keywords: radiation; Tomography, Spiral Computed; Four-Dimensional Computed Tomography; Respiratory Function Tests
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lung Radiation: Patients with tumors in the lung that require radiation therapy

SUMMARY:
It is known that radiation damages lung tissue. New human studies at University of Iowa show that the radiation damage is not as expected. The purpose of this study is to document lung function using four-dimensional computed tomography (CT) and quantify changes three months after radiation therapy for malignant lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of small cell or non-small cell lung cancer or metastatic tumor to the lung being scheduled for localized radiation therapy (including radiosurgery)
* No prior or future planned surgery for the treatment of the lung cancer.
* Age ≥ 18 years
* Karnofsky 60%
* Not pregnant.
* Ability to understand and the willingness to sign a written informed consent document
* Ability and willingness to participate in breathing training and compliance wiht breathing apparatus so that radiation doses are optimally linked to 4D-CT images
* Ability to tolerate CT contrast

Exclusion Criteria:

* No prior thoracic radiotherapy will be permitted
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women
* Severe COPD that requires chronic prednisone or multiple inhalers
* Underlying collagen vascular disease or intrinsic lung disease that could complicate expected sequelae of radiation (idiopathic pulmonary fibrosis, Wegener's granulomatosis)
* Oxygen dependence at baseline
* Recent lung surgery or abdominal surgery (within 3 weeks) that would compromise respiratory pattern.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with lung disease requiring radiation therapy. Lung tumor may be lung cancer or metastasis to the lung. Radiation simulation method must be four-dimensional computer tomography (4D-CT)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-06; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Spirometry correlated to lung expansion maps | 3 months post radiation

CONTACTS AND LOCATIONS:
Overall Officials: John Bayouth, Ph.D., Principal Investigator — University of Iowa; Johm M. Buatti, M.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Department of Radiation Oncology, Iowa City, Iowa, United States